CLINICAL TRIAL: NCT02525536
Title: A Phase 1, Open-Label, Dose Escalation Study Evaluating the Safety, Tolerability and Pharmacokinetics of Trebananib (AMG 386) in Adult Japanese Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study Evaluating the Safety, Tolerability and Pharmacokinetics of Trebananib (AMG 386 ) in Adult Japanese Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060212; U1111-1170-0395 (Registry Identifier: WHO); JapicCTI-101161 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-07-26; First posted 2015-08-17 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-08

CONDITIONS: Neoplasms, Advanced Solid
Keywords: Drug Therapy
MeSH Terms: conditions — Neoplasms | interventions — trebananib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Trebananib 3 mg/kg (Experimental): Trebananib (AMG 386) 3 milligram/kilogram (mg/kg), 60-minute infusion, intravenously once weekly on Days 1, 8, 15 and 22 and thereafter once weekly starting from Day 36 (Week 6) until intolerance to investigational product, progressive disease, consent withdrawn, or lost to follow-up (up to approximately 249 weeks).
  Interventions: Drug: Trebananib 3 mg/kg
- Trebananib 10 mg/kg (Experimental): Trebananib (AMG 386) 10 mg/kg, 60-minute infusion, intravenously once weekly on Days 1, 8, 15 and 22 and thereafter once weekly starting from Day 36 (Week 6) until intolerance to investigational product, progressive disease, consent withdrawn, or lost to follow-up (up to approximately 249 weeks).
  Interventions: Drug: Trebananib 10 mg/kg
- Trebananib 30 mg/kg (Experimental): Trebananib (AMG 386) 30 mg/kg, 60-minute infusion, intravenously once weekly on Days 1, 8, 15 and 22 and thereafter once weekly starting from Day 36 (Week 6) until intolerance to investigational product, progressive disease, consent withdrawn, or lost to follow-up (up to approximately 249 weeks).
  Interventions: Drug: Trebananib 30 mg/kg

INTERVENTIONS:
Drug: Trebananib 3 mg/kg — Trebananib (AMG 386) 3 mg/kg, intravenous infusion.
  Arms: Trebananib 3 mg/kg
Drug: Trebananib 10 mg/kg — Trebananib (AMG 386) 10 mg/kg, intravenous infusion.
  Arms: Trebananib 10 mg/kg
Drug: Trebananib 30 mg/kg — Trebananib (AMG 386) 30 mg/kg, intravenous infusion.
  Arms: Trebananib 30 mg/kg

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetic (PK) profile of trebananib (AMG 386) after intravenous administration in adult Japanese participants with advanced solid tumors.

DETAILED DESCRIPTION:
The drug being tested in this study is called trebananib (AMG 386). Trebananib (AMG 386) is being tested to treat people with advanced solid tumors.

This study will look at the safety, tolerability and pharmacokinetic (PK) profile of trebananib and response to treatment.

The study will enroll approximately 18 participants. Once enrolled, participants will be assigned sequentially into 1 of the 3 cohorts:

* Trebananib 3 milligram/kilogram (mg/kg),
* Trebananib 10 mg/kg,
* Trebananib 30 mg/kg.

All participants will receive trebananib via 60 minute intravenous infusion. This study will be conducted in Japan. The overall time to participate in this study is 14 weeks or more. Participants will attend the end-of-treatment visit 28 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria: 1. Histologically or cytologically documented and definitively diagnosed, advanced solid tumor that is refractory to standard treatment or for which no curative therapy is available. 2. Has Eastern Cooperative Oncology Group (ECOG) of 0 or 1 (within 2 weeks prior to enrollment). 3. Men or women, 20 to 74 years old at the time the written informed consent is obtained. 4. Those meeting the following laboratory criteria (within 2 weeks prior to enrollment): A. Hematological function, as follows: • Absolute neutrophil count >=1500 /microliter (mcL) (without granulocyte colony stimulating factor support within 2 weeks of enrollment). • Platelet count >=10*10^4 /mcL (without transfusion within 2 weeks of enrollment). • Hemoglobin >=9 grams per deciliter (g/dL) (without transfusion within 2 weeks of enrollment). B. Renal function, as follows: • Calculated creatinine clearance (CCr) >40 milliliter per minute (mL/min) according to the Cockcroft-Gault formula. • Urinary protein quantitative value of less than or equal to (<=) 30 mg/dL in urinalysis or <=1+ on dipstick, unless quantitative protein is <=1,000 mg in a 24 hour urine sample. C. Hepatic function, as follows: • AST <=2.5*ULN (if liver metastases are present, <=5*ULN). • ALT <=2.5*ULN (if liver metastases are present, <=5*ULN). • Alkaline phosphatase <=2.0*ULN (if bone or liver metastates present <=5*ULN). • Total bilirubin <=2.0*ULN. D. Hemostatic function, as follows: • Prothrombin time (PT) or activated partial thromboplastin time (APTT) <=1.5*ULN. E. ECG • Normal sinus rhythm (no clinical significant 12-lead ECG changes) 5. Life expectancy of 3 months, in the judgment of the investigator. Exclusion Criteria: 1. Has primary central nervous system (CNS) tumors, including any CNS lymphoma. 2. Has history of CNS metastases (including previously treated metastases) (The brain imaging test by CT or MRI will be performed at screening. If the imaging test was performed within 3 months prior to written informed consent, the result can be used to confirm the exclusion criterion.) 3. Has hematological malignancies. 4. Has unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to CTCAE grade 0 or 1, or to levels specified in the inclusion/exclusion criteria with the exception of alopecia. 5. Has clinically significant cardiovascular disease within 1 year prior to enrollment, including myocardial infarction, unstable angina, New York Heart Association class 2 or greater heart failure, peripheral vascular disease, cerebrovascular accident, transient ischemic attack, or arrhythmias not controlled by outpatient medication. 6. Has uncontrolled hypertension [diastolic >90 millimeter of mercury [mmHg]; systolic >150 mmHg]. Participant on antihypertensive medication must meet these parameters on a stable antihypertensive. 7. Has history of arterial or venous (deep vein) thrombosis within 1 year before enrollment. 8. Has presence of ascites or pleural effusion requiring medical intervention (example, drainage.) 9. Has history of bleeding diathesis or clinically significant bleeding including hemoptysis within 6 months of enrollment. 10. Has non-healing wound, ulcer or fracture. 11. With head and neck cancer. 12. Has squamous cell tumor or lung cancer with large central (located adjacent to or within the hilum or mediastinum) tumor lesions >=3 centimeter (cm), regardless of histology. 13. Has positive test for human immunodeficiency virus infection. 14. Has positive test for hepatitis C virus infection (positive hepatitis C virus antibody [HCVAb] or hepatitis B infection (positive hepatitis B virus antigen [HBsAg] or positive hepatitis B virus antibody [HBcAb])). 15. Had major surgery (requiring general anesthesia) within 4 weeks before enrollment. 16. Has minor surgery, placement of central venous catheter, or fine needle aspiration within 7 days prior to enrollment. 17. Is unable to tolerate IV administration, in the judgment of the investigator. 18. Has prior anti-tumor therapies, defined as: •Treatment with tumor directed antibody therapy within 4 weeks prior to Study Day 1, with the exception of bevacizumab and other monoclonal antibodies with a half-life >10 days, which must be discontinued at least 8 weeks prior to Study Day 1. •Anti-cancer therapy including chemotherapy and retinoid therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin) before Study Day 1. •Hormonal anti-tumor therapy within 4 weeks before Study Day 1. Does not include hormones for non-cancer related conditions (example, insulin for diabetes, hormone replacement therapy). •Therapeutic or palliative radiation therapy within 4 weeks before Study Day 1 (participants must have resolution of any significant adverse effects from radiation therapy received prior to 2 weeks before Study Day 1). 19. Has any elective surgeries scheduled during their participation in the study. 20. Has prior radiation to abdomen. 21. Has concurrent or prior (within 4 weeks before Study Day 1) anticoagulation therapy excluding aspirin and anti-platelet agents. The concurrent use of low molecular weight heparin or low dose warfarin (<=1 mg daily) for prophylaxis against thrombosis is acceptable. 22. Has concurrent immunosuppressant therapy (cyclosporine, tacrolimus, or chronic treatment with prednisolone [> 5 mg daily]) within 4 weeks prior to Study Day 1. 23. Currently or previously treated with angiopoietin inhibitors, or inhibitors of Tie-1 or Tie-2 including, but not limited to, AMG 386, XL880, XL820. 24. Is enrolled in the clinical study for other investigational products or devices or within 4 weeks since the last administration at the enrollment. 25. Is pregnant (example, positive human choriogonadotropin [HCG] test) or breastfeeding. 26. Has a childbearing potential, or participant who has a partner of childbearing potential, who is not using adequate contraceptive precautions, and participant unwilling for 6 months after the last AMG 386 infusion. 27. Has any kind of disorder that compromises the ability of the participant to give written informed consent and/or comply with study procedures. 28. Has any co-morbid medical condition that would increase the risk of toxicity, in the judgement of the investigator or the sponsor. 29. The investigator has determined the participant has difficulties that would prevent the participant's ability to participate in the study. 30. Has a history of allergic reactions to bacterially produced proteins. 31. Has a history of severe drug hypersensitivity.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Result] Doi T, Ohtsu A, Fuse N, Yoshino T, Tahara M, Shibayama K, Takubo T, Weinreich DM. Phase 1 study of trebananib (AMG 386), an angiogenesis targeting angiopoietin-1/2 antagonist, in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2013 Jan;71(1):227-35. doi: 10.1007/s00280-012-2000-1. Epub 2012 Nov 3. PMID 23124648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 26 June 2009 to 28 May 2014.
Pre-assignment Details: Participants with a historical diagnosis of advanced solid tumor were enrolled in 1 of 3 treatment groups: trebananib 3 milligram/kilogram (mg/kg); trebananib 10 mg/kg; trebananib 30 mg/kg.
Groups:
- Trebananib 3 mg/kg: Trebananib (AMG 386) 3 mg/kg, 60-minute infusion, intravenously once weekly on Days 1, 8, 15 and 22 and thereafter once weekly starting from Day 36 (Week 6) until intolerance to investigational product, progressive disease, consent withdrawn, or lost to follow-up (up to approximately 249 weeks).
Period: Overall Study
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all participants who received at least 1 dose of AMG 386.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.41) | 55.3 (7.71) | 60.7 (6.71) | 57.9 (8.22)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 4 | 5 | 3 | 12
  Greater than or equal to (>=) 65 years | 2 | 1 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 4 | 3 | 3 | 10
Height [Mean (Standard Deviation); unit: centimeter] | 162.28 (6.233) | 161.08 (12.788) | 160.48 (3.136) | 161.28 (7.938)
Weight [Mean (Standard Deviation); unit: kilogram] | 52.80 (10.208) | 64.03 (10.623) | 50.40 (3.683) | 55.74 (10.257)
Medical and surgical history [Number; unit: participants]
  With medical and surgical history | 6 | 4 | 5 | 15
  Without medical and surgical history | 0 | 2 | 1 | 3
Primary Tumor Type [Number; unit: participants]
  Neoplasm, stomach | 3 | 0 | 3 | 6
  Neoplasm, rectal | 1 | 2 | 1 | 4
  Neoplasm, pancreatic | 1 | 1 | 1 | 3
  Neoplasm, colon | 1 | 1 | 0 | 2
  Neoplasm, bladder | 0 | 0 | 1 | 1
  Neoplasm, breast | 0 | 1 | 0 | 1
  Neoplasm, uterine | 0 | 1 | 0 | 1
Prior Radiotherapy [Number; unit: participants]
  With prior radiotherapy | 0 | 2 | 0 | 2
  Without prior radiotherapy | 6 | 4 | 6 | 16
Prior Other Cancer Medication [Number; unit: participants]
  With prior other cancer medication | 6 | 6 | 6 | 18
  Without prior other cancer medication | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG Performance status was defined as: 0 = fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (example, light house work, office work); 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Up and about >50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair >50% of waking hours; 4 = completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; or 5 = Dead.
  participants
    ECOG performance status 0 | 6 | 6 | 5 | 17
    ECOG performance status 1 | 0 | 0 | 1 | 1
Method of Tumor Assessment [Number; unit: participants]
  Computed Tomography (CT) | 6 | 6 | 6 | 18
  Magnetic Resonance Imaging (MRI) | 0 | 0 | 0 | 0
Number of Target Lesions [Number; unit: participants]
  1 Target Lesion | 0 | 1 | 1 | 2
  2 Target Lesion | 2 | 0 | 2 | 4
  3 Target Lesion | 2 | 0 | 0 | 2
  4 Target Lesion | 0 | 0 | 2 | 2
  >=5 Target Lesion | 2 | 5 | 1 | 8
Sum of the Longest Diameter of Target Lesions [Mean (Standard Deviation); unit: millimeters] | 112.3 (98.70) | 179.3 (99.23) | 96.8 (63.07) | 129.5 (91.04)
Presence of Non-Target Lesions [Number; unit: participants]
  With Non-Target Lesions | 6 | 6 | 6 | 18
  Without Non-Target Lesions | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Enrollment in Japan is reported in this measure.
  participants | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT is defined as any treatment-related, grade 4 or higher hematologic or grade 3 or higher non-hematologic toxicity (according to the Common Terminology Criteria for Adverse Events [CTCAE] version 3.0; hematologic toxicity means any toxicities which are categorized in blood/bone marrow category of CTCAE), except for aspartate aminotransferase (AST), alanine aminotransferase (ALT) and infusion reaction, occurred during the first 28 days after the initial administration (before examination on Study Day 29). DLT also includes AST or ALT: >10*upper limit of normal (ULN) international units per liter (IU/L).
Time Frame: Day 1 up to Day 28
Population: DLT analysis set: all participants who experience at least 1 DLT in the first 28 days of treatment, or who received all planned AMG 386 dose and are followed until the day before the treatment on Study Day 29.
Measure: Number; unit: participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (AEs) and Serious Adverse Event (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. Treatment emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: Baseline up to 4 weeks after the last dose of study drug, where last dose was given up to Week 249
Population: Safety analysis set: all participants who received at least 1 dose of AMG 386.
Measure: Number; unit: participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants
  AEs | 6 | 6 | 6
  SAEs | 2 | 0 | 1

3. Primary Outcome: Number of Participants With Significant Change From Baseline in Electrocardiogram (ECG)
Description: Change relative to baseline in electrocardiogram measured throughout study. Significant change in ECG observed at any time point was summarized and reported.
Time Frame: Week 1: predose, 1, 6 hours after end of infusion, Week 4: predose, 1 hour after end of infusion, Week 8, 16: predose, thereafter predose of every 8 weeks up to 4 weeks after the last dose of study drug, where last dose was given up to Week 249
Population: Safety analysis set: all participants who received at least 1 dose of AMG 386.
Measure: Number; unit: participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature, diastolic and systolic blood pressure, and pulse (beats per minutes). clinically significant change in vital signs observed at any time point was summarized and reported.
Time Frame: Week 1: predose, 1, 2, 6, 24, 48 and 96 hours after infusion end, Week 2, 3, 4: predose and 1 hour after infusion end, thereafter predose of every 4 weeks starting from Week 8 up to 4 weeks after the last dose of study drug (last dose=Week 249)
Population: Safety analysis set: all participants who received at least 1 dose of AMG 386.
Measure: Number; unit: participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Laboratory Values
Description: The number of participants with any abnormal standard safety laboratory values collected throughout study. Parameters assessed were hematology, chemistry, coagulation and urinalysis. Abnormal laboratory values observed at any time point was summarized and reported.
Time Frame: Week 1: predose, 24, 48 and 96 hours after infusion end, Week 2 and 3: predose, Week 4: predose and 1 hour after infusion end, thereafter every 4 weeks starting from Week 8 up to 4 weeks after the last dose of study drug (last dose=Week 249)
Population: Safety analysis set: all participants who received at least 1 dose of AMG 386.
Measure: Number; unit: participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants
  Hematology | 5 | 4 | 6
  Chemistry | 6 | 6 | 6
  Coagulation | 3 | 0 | 0
  Urinalysis | 2 | 2 | 3

6. Primary Outcome: Cmax: Maximum Observed Serum Concentration for AMG 386 After Week 1 Dose
Description: Maximum observed serum concentration (Cmax) is the peak serum concentration of a drug after administration, obtained directly from the serum concentration-time curve.
Time Frame: Week 1: predose, 1, 2, 6, 24, 48 and 96 hours after end of infusion, Week 2: predose
Population: Pharmacokinetic analysis set: all participants who had at least 1 evaluable serum concentrations, received at least 1 dose of AMG 386, and had Week 1 assessment available.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
microgram per milliliter (mcg/mL) | 52.33 (11.27) | 239.0 (47.11) | 551.2 (86.76)

7. Primary Outcome: Cmax: Maximum Observed Serum Concentration for AMG 386 After Week 4 Dose
Description: Cmax is the peak serum concentration of a drug after administration, obtained directly from the serum concentration-time curve.
Time Frame: Week 4: predose, 1, 2, 6, 24, 48, 96, 168 and 264 hours after end of infusion
Population: Pharmacokinetic analysis set: all participants who had at least 1 evaluable serum concentrations, received at least 1 dose of AMG 386, and had Week 4 assessment available.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
mcg/mL | 59.02 (10.09) | 277.0 (48.79) | 688.7 (104.5)

8. Primary Outcome: Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for AMG 386 After Week 1 Dose
Description: Tmax is the time to reach the maximum serum concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Week 1: predose, 1, 2, 6, 24, 48 and 96 hours after end of infusion, Week 2: predose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
hour (hr) | 1.067 (582.1) [1.033 to 1.083] | 1.033 (924.5) [1.017 to 1.050] | 1.167 (4489) [1.017 to 2.000]

9. Primary Outcome: Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for AMG 386 After Week 4 Dose
Description: Tmax is the time to reach the maximum serum concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Week 4: predose, 1, 2, 6, 24, 48, 96, 168 and 264 hours after end of infusion
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
hr | 1.067 (35.05) [1.017 to 2.033] | 1.017 (14.84) [1.017 to 2.017] | 1.508 (25.57) [1.033 to 2.017]

10. Secondary Outcome: Number of Participants With Best Overall Response
Description: Best overall response for a participant is the best observed post-baseline disease response as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 criteria. Complete Response (CR): disappearance of all target lesions, non-target lesions and normalization of tumor marker level. Partial Response (PR): at least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the baseline smallest sum of longest diameter; persistence of 1 or more non-target lesion(s) or maintenance of tumor marker level above the normal limits. PD: at least 20% increase in the sum of the longest diameter of target lesions, taking as reference the baseline smallest sum of longest diameter or appearance of 1 or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Baseline, assessed every 8 weeks up to 4 weeks after the last dose of study drug, where last dose was given up to Week 249
Population: Response evaluable analysis set: a subset of participants in the full analysis set (FAS) with at least 1 measurable lesion at baseline using the RECIST 1.0. FAS consisted of all participants who had evaluable data and received at least 1 dose of AMG 386.
Measure: Number; unit: participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants
  CR | 0 | 0 | 0
  PR | 1 | 0 | 1
  SD | 0 | 1 | 1
  PD | 5 | 5 | 4

11. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response rate defined as the rate of participants with CR or PR based on RECIST 1.0 criteria. CR: disappearance of all target lesions, non-target lesions and normalization of tumor marker level. PR: at least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: as for outcome 10
Population: Response evaluable analysis set: a subset of participants in the FAS with at least 1 measurable lesion at baseline using the RECIST 1.0. FAS consisted of all participants who had evaluable data and received at least 1 dose of AMG 386.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Percentage of participants | 17 [0.4 to 64.1] | 0 [0.0 to 39.3] | 17 [0.4 to 64.1]

12. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of first administration of study treatment to the date of first documentation of PD or death caused by progression. For participants who did not have a documented PD or died owing to causes other than progression, TTP was censored at the time of last response assessment. PD is defined as at least 20% increase in the sum of the longest diameter of target lesions, taking as reference the baseline smallest sum of longest diameter or appearance of 1 or more new lesions or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 10
Population: Response evaluable analysis set: a subset of participants in the FAS with at least 1 measurable lesion at baseline using the RECIST 1.0. FAS consisted of all participants who had evaluable data and received at least 1 dose of AMG386.
Measure: Median (Full Range); unit: Days
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Days | 48.0 [26 to 1221] | 46.0 [15 to 150] | 45.5 [45 to 718]

13. Secondary Outcome: Percent Change From Baseline to Post-baseline in the Sum of the Longest Diameters of Tumor
Description: The percent change from baseline to post-baseline is the largest percent reduction from baseline among all post-dose measures of the sum of the longest diameter of the tumor burden.
Time Frame: as for outcome 10
Population: Response evaluable analysis set: a subset of participants in the FAS with at least 1 measurable lesion at baseline using the RECIST 1.0 and valid post-baseline tumor lesion assessment available. FAS consisted of all participants who had evaluable data and received at least 1 dose of AMG 386.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 5 | 6 | 6
percent change | -1.53 (48.655) | 16.36 (18.455) | 5.53 (46.907)

14. Secondary Outcome: Number of Participant With Anti-AMG 386 Antibody
Description: The immunogenicity of AMG 386 was evaluated with an immunoassay that detects anti-AMG 386 binding antibodies. Antibody formation reported at any of the time points was summarized.
Time Frame: Week 1: predose,1,2,6,24,48 and 98 hours after infusion end, Week 3: predose, Week 4: predose, 1,2,6,24,48,96,168 and 264 hours after infusion end, thereafter predose every 4 weeks starting from Week 8 up to 8 weeks after last dose (last dose=Week 249)
Population: Safety analysis set: all participants who received at least 1 dose of AMG 386.
Measure: Number; unit: participants
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
participants | 2 | 1 | 0

15. Primary Outcome: AUC (0-tau): Area Under the Serum Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for AMG 386 After Week 1 Dose
Description: AUC (0-tau) is the area under the serum concentration-time curve during a dosing interval, where tau is the length of the dosing interval (168 hours for once weekly regimen).
Time Frame: Week 1: predose, 1, 2, 6, 24, 48 and 96 hours after end of infusion, Week 2: predose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microgram*hour/milliliter (mcg*hr/mL)
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
microgram*hour/milliliter (mcg*hr/mL) | 1760 (582.1) | 4629 (924.5) | 18040 (4489)

16. Primary Outcome: AUC (0-tau): Area Under the Serum Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for AMG 386 After Week 4 Dose
Description: as for outcome 15
Time Frame: Week 4: predose, 1, 2, 6, 24, 48, 96, and 168 hours after end of infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
mcg*hr/mL | 2171 (715.4) | 5880 (559.6) | 21170 (2912)

17. Primary Outcome: Cmin: Minimum Observed Serum Trough Concentration for AMG 386 After Week 1 Dose
Description: Cmin was the observed serum concentration at 168 hours postdose.
Time Frame: Week 2: predose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
mcg/mL | 2.702 (1.226) | 3.857 (1.018) | 20.20 (5.060)

18. Primary Outcome: Cmin: Minimum Observed Serum Trough Concentration for AMG 386 After Week 4 Dose
Description: Cmin was the observed serum concentration at 168 hours postdose.
Time Frame: Week 4: 168 hours after end of infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
mcg/mL | 5.323 (2.536) | 7.266 (1.521) | 45.07 (16.24)

19. Primary Outcome: Vss: Volume of Distribution at Steady State for AMG 386
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state, estimated as: Vss = MRTinf *CLss, where MRTinf is mean residence time of drug extrapolated to infinity and CLss is the systemic clearance at the steady state. Vss was normalized to participant's body weight.
Time Frame: Week 4: predose, 1, 2, 6, 24, 48, 96, 168 and 264 hours after end of infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
milliliter per kilogram (mL/kg) | 158.2 (49.02) | 121.0 (22.18) | 136.6 (30.26)

20. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for AMG 386
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Time Frame: Week 4: predose, 1, 2, 6, 24, 48, 96, 168 and 264 hours after end of infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
hr | 95.86 (35.05) | 95.41 (14.84) | 93.89 (25.57)

21. Primary Outcome: Systemic Clearance at Steady State (CLss) for AMG 386
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. Systemic clearance at steady state (CLss) was calculated as the ratio of dose administered to AUC (0 - tau), where AUC (0 - tau) is the area under the serum concentration-time curve during a dosing interval, where tau is the length of the dosing interval (168 hours for once weekly regimen). CLss was normalized to participant's body weight.
Time Frame: Week 4: predose, 1, 2, 6, 24, 48, 96 and 168 hours after end of infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliter/hour/kilogram(mL/hr/kg)
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
milliliter/hour/kilogram(mL/hr/kg) | 1.495 (0.4231) | 1.713 (0.1653) | 1.439 (0.1912)

22. Primary Outcome: Accumulation Ratio (AR) for AMG 386
Description: Accumulation ratio (AR) was calculated by dividing the individual AUC (0-tau) value at Week 4 by the corresponding individual AUC (0-tau) value at Week 1.
Time Frame: Week 1: predose, 1, 2, 6, 24, 48 and 96 hours after end of infusion, Week 2: predose, Week 4: predose, 1, 2, 6, 24, 48, 96, and 168 hours after end of infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Number analyzed (Participants) | 6 | 5 | 6
ratio | 1.235 (0.05143) | 1.193 (0.06862) | 1.211 (0.2139)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of the study drug and no more than 28 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Trebananib 3 mg/kg | Trebananib 10 mg/kg | Trebananib 30 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trebananib 3 mg/kg (N=6) | Trebananib 10 mg/kg (N=6) | Trebananib 30 mg/kg (N=6)
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trebananib 3 mg/kg (N=6) | Trebananib 10 mg/kg (N=6) | Trebananib 30 mg/kg (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Corneal erosion (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 2 | 3
Fatigue (General disorders) | 3 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 2
Influenza like illness (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0
Ovarian infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 3 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.